CLINICAL TRIAL: NCT06887959
Title: A Phase 4, Open-label, Single-arm Study Evaluating the Effectiveness and Safety of Suzetrigine As Part of Multimodal Therapy for Acute Pain After Laparoscopic Procedures of the Intraperitoneal or Retroperitoneal Cavities or Arthroscopic Orthopedic Procedures
Brief Title: A Single-arm Study Evaluating the Effectiveness and Safety of Suzetrigine (SUZ) for Acute Pain After Selected Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-548-108
Record Dates: First submitted 2025-03-19; First posted 2025-03-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Suzetrigine (SUZ) (Experimental): Participants will receive SUZ for 14 days or until their pain resolves, whichever occurs first.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ; Journavx

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and tolerability of SUZ for acute pain after laparoscopic procedures of the intraperitoneal or retroperitoneal cavities or arthroscopic orthopedic procedures.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of greater than or equal to (≥) 18.0 to less than or equal to (≤) 40.0 kilogram per meter square (kg/m^2)
* Scheduled to undergo a procedure that is in one of the following categories that would typically be treated with opioid therapy for at least 72 hours postoperatively such as

  * Laparoscopic intraperitoneal or retroperitoneal procedure
  * Arthroscopic orthopedic procedure

Key Exclusion Criteria:

-Participated in previous study with Suzetrigine or received Journavx

Other protocol defined Inclusion/Exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Reporting Good, Very Good, or Excellent on a Patient Global Assessment (PGA) for Pain Control at the End of Treatment | From Day 3 up to Day 14

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Gulfcoast Research Institute, Sarasota, Florida
  - MedStar, Baltimore, Maryland
  - Oasis Clinical Research, Las Vegas, Nevada
  - Cooper University HealthCare (CUH), Camden, New Jersey
  - North Shore University Hospital - Anesthesiology, Manhasset, New York
  - OrthoCarolina - Hip & Knee Center, Charlotte, North Carolina
  - Eximia Research-Durham, Durham, North Carolina
  - Duke University Hospital - Anesthesiology, Durham, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Seaside Clinical Research Institute, Wilmington, North Carolina
  - UH Cleveland Medical Center - Anesthesiology, Cleveland, Ohio
  - University of Tennessee Medical Center - Anethesiology, Knoxville, Tennessee
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - Memorial Hermann Village, Houston, Texas
  - Tidewater Clinical Research, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/